CLINICAL TRIAL: NCT07147608
Title: Simplification of PHysical Activity Assessment by Rapid Interrogation - Phase 2
Brief Title: SAPHIR2 : Simplification of PHysical Activity Assessment by Rapid Interrogation
Acronym: SAPHIR2
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC25_0220
Record Dates: First submitted 2025-08-21; First posted 2025-08-29 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: General Population (no Specific Condition or Disease)
Keywords: exercise; sedentary behavior; sports medicine
MeSH Terms: conditions — Disease; Motor Activity; Sedentary Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SAPHIR2 cohort: Initial physical activity questionnaire, wearing the actimeter for 7 days, final physical activity questionnaire
  Interventions: Other: actimeter wearing; Other: physical activities questionnaires

INTERVENTIONS:
Other: actimeter wearing — actimeter wearing during 7 days : recording of physical activity over 7 days using a non-invasive external sensor
Other: physical activities questionnaires — IPAQ and SAPHIR questionnaires

SUMMARY:
A multicentric, non-interventional study using a clinical questionnaire (SAPHIR) and activity monitor (Activ-PAL) to estimate the level of physical activity in the general population.

This study compares the level of physical activity reported by the SAPHIR questionnaire with the activity recorded by the activity monitor during the same period, in order to determine if the SAPHIR score is able to represent the measured physical activity, in a simple and easily calculable manner.

Hypothesis:

The aim of this work is to propose a new questionnaire that is simple to complete by the patient,quick to analyse and directly calculable by the doctor and adapted to the general population, whether during the initial evaluation or the follow-up.

Indeed, these scores are rarely used outside the context of the prescription of physical activity in specialized centers. Moreover, a tool suited to the constraints of community medicine seems necessary, given the growth of the prescription of physical activity in primary care.

The idea behind this new questionnaire is to obtain a score ranging from 0 to 100 that can be calculated through simple mental arithmetic, which is not the case for most existing questionnaires, in particular the IPAQ.

DETAILED DESCRIPTION:
Promotion of physical activity has been an important public health issue in France for around ten years, as demonstrated by numerous reports and public health plans 'qui ont vu le jour" with this aim. (Plan national nutrition santé PNNS 2011-2015 ; Plan obésité PO 2010-2013 ; Plan cancer 2014-2019). In order to continue promoting physical activity (PA), it is necessary to have a well-adapted, simple and rapid tool is that allows precise evaluation and monitoring within the general population.

Currently, the French National Authority for Health (la Haute Autorité de Santé), through its guide for the promotion, consultation and medical prescription of physical and sports activity for health in adults, updated in July 2022, proposes an estimate of the "usual level of PA (…) using the two-question Marshall questionnaire (30 seconds)" or alternatively, "it can be calculated more precisely with the Global Physical Activity Questionnaire (GPAQ), a 16-question self-administered questionnaire that patients can complete online at www.mangerbouger.fr."

The GPAQ is one of the most widely used questionnaires. While its strength lies in its precision, it is long to complete and score. Therefore, despite being validated by many studies, it is not practical for routine use. In practice, the "Ricci and Gagnon" questionnaire is used for the follow-up of patients, using tracking logs. (Sport santé sur ordonnance. Contexte et exemples de mise en oeuvre. Octobre 2017. ONAPS) . This categorizes individuals as inactive, active or very active, and has never been scientifically validated in a study, to the best of our knowledge.

Finally, the International Physical Activity Questionnaire (IPAQ) is a test validated both in long and short forms. It allows a precise calculation of the amount of physical activity expressed in MET (metabolic equivalent)/min/week but does not provide information on its distribution throughout the week. Like the GPAQ, with 27 different questions it is also lengthy to complete, making it impractical for routine use. The short version tends to underestimate physical activity levels, and the final score cannot be easily calculated in real time. Nevertheless, this version will be used as a reference.

The aim of this work is to propose a new questionnaire that is simple for patients to complete, quick to analyse, can be calculated directly by the doctor, and is adapted to the general population, whether for an initial assessment or a follow-up.

Moreover, the prescription of physical activity is usually carried out over short, renewable periods, whereas long-term changes are necessary to achieve significant improvements in morbidity and mortality.

The developed questionnaire ultimately aims to be useful for monitoring the evolution of physical activity.

ELIGIBILITY:
Inclusion criteria:

* Patients referred for a consultation at one of the participating centers
* Patients over 18 years old with no upper age limit

Non-inclusion criteria:

* Patients with a contra-indication to walking
* Professional athletes or patients participating in endurance sports competitions
* Patients refusing to participate in the study
* Patients unable to understand the objectives or instructions of the study

Exclusion criteria:

-Patients with Activ-PAL recordings of less than 3 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consists of patients referred for consultation in the department of sports medicine (generally active patients, although patients may also be sedentary and/or inactive) or in the department of vascular medicine (patients with lower limb peripheral artery disease, mostly inactive)
Sampling Method: Non-Probability Sample
Enrollment: 118 (Estimated)
Dates: Start 2025-12-19 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
correlation between SAPHIR score completed at inclusion and the level of physical activity estimated from measurement data collected using the Activ-PAL® activity monitor | 7 days
  A score is based on the time spent at each intensity level of physical activity, using the correlation between cadence and METs extrapolated from the literature (Tudor-Locke et al, 2020). The primary outcome measure is the correlation coefficient between the amount of physical activity estimated by the SAPHIR score and that estimated from the Activ-PAL data.

SECONDARY OUTCOMES:
correlation between the final SAPHIR score (completed at the end of the measurement week) and the amount of physical activity calculated from the Activ-PAL® activity monitor data | 7 days
  The first secondary outcome measure is the correlation coefficient between the SAPHIR score and the amount of activity estimated from Activ-PAL® data.
correlation between the initial SAPHIR score and the IPAQ score (baseline) | inclusion
  The second secondary outcome measure is the correlation coefficient between the initial SAPHIR score and the initial IPAQ score
correlation between the final SAPHIR score and the final IPAQ score | 7 days
  The third secondary outcome measure is the correlation coefficient between the final SAPHIR score and the final IPAQ score
correlation between the initial IPAQ score (at the beginning of the week) and the amount of physical activity calculated using Activ-PAL® data i | 7 days
  The fourth secondary outcome measure is the correlation coefficient between the initial IPAQ score and the amount of physical activity estimated from Activ-PAL® data, using the method described for the primary outcome
correlation between the final IPAQ score (at the end of the recording week) and the amount of physical activity calculated using Activ-PAL® data | 7 days
  The fifth secondary outcome measure is the correlation coefficient between the final IPAQ score and the amount of activity measured from Activ-PAL® data, following the method described for the primary outcome

CONTACTS AND LOCATIONS:
Overall Officials: Simon LECOQ, MD, Principal Investigator — University Hospital, Angers
Locations (3):
- France (3):
  - CHU d'Angers, Angers
  - CH de Cholet, Cholet
  - CH du Mans, Le Mans

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hillsdon M, Foster C, Thorogood M. Interventions for promoting physical activity. Cochrane Database Syst Rev. 2005 Jan 25;2005(1):CD003180. doi: 10.1002/14651858.CD003180.pub2. PMID 15674903
- [Result] Kwak L, Hagstromer M, Sjostrom M. Can the IPAQ-long be used to assess occupational physical activity? J Phys Act Health. 2012 Nov;9(8):1130-7. doi: 10.1123/jpah.9.8.1130. Epub 2011 Dec 27. PMID 22207150
- [Result] Joseph KL, Dagfinrud H, Christie A, Hagen KB, Tveter AT. Criterion validity of The International Physical Activity Questionnaire-Short Form (IPAQ-SF) for use in clinical practice in patients with osteoarthritis. BMC Musculoskelet Disord. 2021 Feb 27;22(1):232. doi: 10.1186/s12891-021-04069-z. PMID 33639913
- [Result] Curry WB, Thompson JL. Comparability of accelerometer- and IPAQ-derived physical activity and sedentary time in South Asian women: A cross-sectional study. Eur J Sport Sci. 2015;15(7):655-62. doi: 10.1080/17461391.2014.957728. Epub 2014 Sep 24. PMID 25252088
- [Result] Wu Y, Johns JA, Poitras J, Kimmerly DS, O'Brien MW. Improving the criterion validity of the activPAL in determining physical activity intensity during laboratory and free-living conditions. J Sports Sci. 2021 Apr;39(7):826-834. doi: 10.1080/02640414.2020.1847503. Epub 2020 Nov 18. PMID 33203323
- [Result] Tudor-Locke C, Aguiar EJ, Han H, Ducharme SW, Schuna JM Jr, Barreira TV, Moore CC, Busa MA, Lim J, Sirard JR, Chipkin SR, Staudenmayer J. Walking cadence (steps/min) and intensity in 21-40 year olds: CADENCE-adults. Int J Behav Nutr Phys Act. 2019 Jan 17;16(1):8. doi: 10.1186/s12966-019-0769-6. PMID 30654810
- [Result] Tudor-Locke C, Ducharme SW, Aguiar EJ, Schuna JM Jr, Barreira TV, Moore CC, Chase CJ, Gould ZR, Amalbert-Birriel MA, Mora-Gonzalez J, Chipkin SR, Staudenmayer J. Walking cadence (steps/min) and intensity in 41 to 60-year-old adults: the CADENCE-adults study. Int J Behav Nutr Phys Act. 2020 Nov 10;17(1):137. doi: 10.1186/s12966-020-01045-z. PMID 33168018